CLINICAL TRIAL: NCT00549848
Title: Total Therapy Study XVI for Newly Diagnosed Patients With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Enzon Pharmaceuticals, Inc. (Industry); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOTXVI; R01CA140729 (NIH); F32CA141762 (NIH); R37CA036401 (NIH); R01CA090246 (NIH); Aspar PK-PD-T16 (Other: Enzon Pharmaceuticals, Inc.); NCI-2011-01254 (Registry Identifier: NCI Clinical Trial Registration Program); P50GM115279 (NIH)
Record Dates: First submitted 2007-10-25; First posted 2007-10-26 (Estimated); Results first posted 2022-02-10 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-07

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Prednisone; Vincristine; Daunorubicin; pegaspargase; asparaginase erwinia chrysanthemi recombinant; Doxorubicin; Cyclophosphamide; Cytarabine; Thioguanine; 6-thioguanylic acid; Clofarabine; Methotrexate; Mercaptopurine; Dexamethasone; Etoposide; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HD PEG (Experimental): Participants randomized to receive higher dose PEG-asparaginase during the continuation phase.
  Interventions:
  * Prednisone, Vincristine, Daunorubicin, PEG-L-asparaginase, Erwinia L-asparaginase, Doxorubicin, Cyclophosphamide, Cytarabine, Thioguanine
  * Clofarabine, Methotrexate, Mercaptopurine, Dexamethasone, Etoposide, Dasatinib
  Interventions: Drug: Prednisone, Vincristine, Daunorubicin, PEG-L-asparaginase, Erwinia L-asparaginase, Doxorubicin, Cyclophosphamide, Cytarabine, Thioguanine; Drug: Clofarabine, Methotrexate, Mercaptopurine, Dexamethasone, Etoposide, Dasatinib
- CD PEG (Active Comparator): Participants randomized to receive conventional dose PEG-asparaginase during the continuation phase..
  Interventions:
  * Prednisone, Vincristine, Daunorubicin, PEG-L-asparaginase, Erwinia L-asparaginase, Doxorubicin, Cyclophosphamide, Cytarabine, Thioguanine
  * Clofarabine, Methotrexate, Mercaptopurine, Dexamethasone, Etoposide, Dasatinib
  Interventions: Drug: Prednisone, Vincristine, Daunorubicin, PEG-L-asparaginase, Erwinia L-asparaginase, Doxorubicin, Cyclophosphamide, Cytarabine, Thioguanine; Drug: Clofarabine, Methotrexate, Mercaptopurine, Dexamethasone, Etoposide, Dasatinib

INTERVENTIONS:
Drug: Prednisone, Vincristine, Daunorubicin, PEG-L-asparaginase, Erwinia L-asparaginase, Doxorubicin, Cyclophosphamide, Cytarabine, Thioguanine — See Detailed Description section for details of treatment interventions.
  Other Names: Prednisone: prednisolone; Vincristine: Oncovin(R); Daunorubicin: daunomycin, Cerubidine(R); PEG-L-asparaginase: pegaspargase, Oncaspar(R); Erwinia L-Asparaginase: Erwinase(R); Doxorubicin: Adriamycin(R); Cyclophosphamide: Cytoxan(R); Cytarabine: Ara-C, Cytosar-U(R); Thioguanine: 6-TG
Drug: Clofarabine, Methotrexate, Mercaptopurine, Dexamethasone, Etoposide, Dasatinib — See Detailed Description section for details of treatment interventions.
  Other Names: Clofarabine: clofarex, Clolar(TM); Methotrexate: MTX; Mercaptopurine: 6-MP, Purinethol(R); Dexamethasone: Decadron(R); Etoposide: VP-16, Vepesid(R); Dasatinib: Sprycel(R)

SUMMARY:
The primary objective of this study (TOTXVI) is to compare the clinical benefit, the pharmacokinetics, and the pharmacodynamics of polyethylene glycol-conjugated (PEG) asparaginase given in higher dose (HD PEG) versus those of PEG-asparaginase given in conventional dose (CD PEG) during the continuation phase.

This study has several secondary objectives:

Therapeutic Objectives:

To estimate the event-free survival and overall survival of children with ALL who are treated with risk-directed therapy.

To study whether intensifying induction, including fractionated cyclophosphamide and thioguanine, in patients with day 15 MRD > 5%, will result in improved leukemia cytoreduction in this subgroup compared to TOTXV.

To assess whether intensification of central nervous system (CNS)-directed intrathecal and systemic chemotherapy will improve outcome in patients at high risk of CNS relapse.

Exploratory Pharmacologic Objectives:

To identify pharmacogenetic, pharmacokinetic and pharmacodynamic predictors for treatment-related outcomes in the context of the systemic therapy used in the protocol.

To compare the pharmacokinetics and pharmacodynamics of PEG-asparaginase given in higher dose (3,500 or 3,000 units/m2) versus those of PEG-asparaginase given in conventional dose (2,500 units/m2) in the continuation phase.

Exploratory Biologic Objectives:

To determine the prognostic value of levels of minimal residual disease in peripheral blood at day 8 of remission induction.

To validate new markers and methods for MRD detection. To genotype natural killer (NK) cell receptors and measure their expressions at diagnosis and before reinduction, and to associate these features with treatment outcome.

To identify new prognostic factors by applying new technologies to study patient material (e.g., stored plasma, serum, cerebrospinal fluid, and normal and leukemic cells).

Exploratory Neuroimaging Objectives:

To use quantitative MR measures (Diffusion Tensor Imaging and high resolution volumetric imaging) to assess differences in myelin and cortical thickness development in patients treated for ALL relative to healthy controls matched for age and gender.

To assess the impact of folate pathway genetic polymorphisms on myelin and cortical thickness development and neurocognitive performance.

To assess the impact of frontal-parietal lobe myelin and cortical thickness development on neurocognitive performance in attention, working memory, fluency, visual-spatial reasoning and processing speed.

DETAILED DESCRIPTION:
Details of the Treatment Plan:

Treatment will consist of three main phases: Remission Induction, Consolidation, and Continuation.

1. Remission Induction

   * Intrathecal Treatment during Induction

   Frequency and total number of triple intrathecal treatments for Remission Induction is based on the patient's risk of CNS relapse.All patients will receive triple intrathecal treatment on days 1 and 15. Patients with high risk features may receive additional triple intrathecal treatment on days 4, 8, 11, and 22.[t(1;19)/E2A-PBX1.

   Induction treatment will begin with prednisone, vincristine, daunorubicin, PEG-asparaginase and triple intrathecal treatment, followed by cyclophosphamide plus cytarabine plus thioguanine.

   Remission Induction Chemotherapy (6-7 weeks) Prednisone 40 mg/m2/day PO (divided t.i.d.) Days 1 - 28 Dexamethasone will be substituted for prednisone in patients with early T-cell precursor (ETP) immunophenotype.

   Mercaptopurine will be substituted for thiopurine in TPMT HET/deficient patients Dexamethasone (for ETP immunophenotype only) 10 mg/m2/day PO (divided t.i.d.)Days 1-21; 4 mg/m2/day PO (divided t.i.d) Days 22-24; 2 mg/m2/day PO(divided t.i.d) Days 25-28 Vincristine 1.5 mg/m2 IV (max 2 mg) Days 1, 8, 15, 22 Daunorubicin 25 mg/m2 IV Days 1 and 8 PEG-asparaginase 3,000 Units/m2 IV Day 3

   - Participants with Day 15 MRD greater than or equal to 1%: PEG-asparaginase 3,000 Units/m2 IV Day 15

   - Participants with Day 15 MRD less than 5% (excluding MLL positive infants): Cyclophosphamide 1000 mg/m2 IV Day 22 Cytarabine 75 mg/m2/dose IV Days 23-26, 30-33 Thioguanine [Mercaptopurine (TPMT HET/deficient patients only)]60 mg/m2/dose PO Days 22-35 Dasatinib (Ph+ participants only) 40 mg/m2 b.i.d starting Day 22 of induction to continue until end of treatment

   Day 15 MRD > or equal to 5% (excluding MLL+ infants) Cyclophosphamide† 300 mg/m2 IV/ q12 hrs on Days 22-23 Cytarabine 75 mg/m2/dose IV Days 23-26, 30-33 Thioguanine [Mercaptopurine (TPMT HET/deficient patients only) 60 mg/m2/dose PO Days 22-35 Dasatinib‡ (Ph+ participants only) 40 mg/m2 b.i.d Daily Starting Day 22 of induction to continue until end of treatment

   - Infants with MLL positive rearrangement: Clofarabine 40 mg/m2/dose IV Days 22-26 Etoposide 100 mg/m2/dose IV Days 22-26 Cyclophosphamide 300 mg/m2/dose IV Days 22-26
2. Consolidation Treatment (8 weeks) High Dose Methotrexate (HDMTX) 2.5 gm/ (low risk), or targeted 65 μM (std/high-risk) days 1, 15, 29 and 43. Mercaptopurine 50 mg/m2/day Days 1 to 56. All patients will receive triple intrathecal therapy every other week for four doses on Days 1, 15, 29, and 43. Dose is age dependent.

   - Reintensification

   Patients with high-risk leukemia may receive reintensification therapy and then will be offered the option of transplant. This treatment will attempt to maximize leukemic cell kill before allogeneic hematopoietic stem cell transplantation.

   Dexamethasone 20 mg/m2/day PO or IV Days 1-6.Cytarabine 2 grams/m2, 3-hour IV infusion every 12 hours Days 1-2. Etoposide 100 mg/m2, 1-hour IV infusion every 12 hours Days 3-5. Intrathecal methotrexate+hydrocortisone+cytarabine (ITMHA) Day 5; PEG-asparaginase 3,000 units/m2 IV Day 6

   Patients with suboptimal response to reintensification may receive one to two cycles of clofarabine/cyclophosphamide/etoposide/dexamethasone:

   Clofarabine 40 mg/m2/day, 2-hour IV infusion Days 1-5 Etoposide 100 mg/m2/day, 2-hour IV infusion Days 1-5 Cyclophosphamide 300 mg/m2/day, 30-60 minute IV infusion Days 1-5 Dexamethasone 8 mg/m2/day (divided t.i.d) Days 1-5
3. Continuation Treatment (120 weeks)

Abbreviations used below: DEX=dexamethasone; DOX=doxorubicin; VCR=vincristine; MP=mercaptopurine; PEG-ASP=polyethylene glycol-conjugated asparaginase; MTX=methotrexate; 6MP=mercaptopurine

Weeks 1 through 20 - treatment depends on risk assignment standard-high versus low-risk

Week Standard-/High-Risk Low-Risk

1. DEX+DOX+VCR+MP + PEG-ASP/MP + DEX + VCR
2. MP MP + MTX
3. MP + PEG-ASP/MP + MTX
4. DEX + DOX + VCR + MP/MP + DEX + VCR
5. MP + PEG-ASP MP + MTX
6. MP MP + MTX
7. Reinduction I
8. Reinduction I
9. Reinduction I
10. MP/MP + MTX
11. DOX + VCR +MP + PEG-ASP/MP + MTX
12. MP/MP + MTX
13. MP + PEG-ASP/MP + MTX
14. DEX + DOX + VCR +6MP/MP + DEX + VCR
15. MP + PEG-ASP/MP + MTX
16. MP/MP + MTX
17. Reinduction II
18. Reinduction II
19. Reinduction II
20. No chemotherapy/MP + MTX

    Drug Dosages, Schedules and Routes for Continuation Therapy Weeks 1 to 6 and 10 to 16:

    Dexamethasone 12 mg/m2 (std/high risk) or 8 mg/m2 (low risk) PO daily (divided t.i.d.) for 5 days, Days 1-5. Doxorubicin 30 mg/m2 IV, Day 1. Vincristine 2 mg/m2 IV push (max. 2 mg), Day 1 (0.05 mg/kg for patients < 1 year of age or < 10kg in weight). MP (mercaptopurine) 50 mg/m2 PO daily for 7 days (std/high risk), Days 1-7, 75 mg/m2 PO daily for 7 days (low risk), Days 1-7. PEG-ASP (PEG-asparaginase) 2,500 vs. 3,500 units/m2 IV randomization, Day 1. Methotrexate 40 mg/m2 IV Day 1.

    Dexamethasone, vincristine, and asparaginase will be given regardless of blood counts, provided that the patient is clinically well. Doxorubicin, mercaptopurine and methotrexate will be held if white blood count (WBC) <1000/mm3 or absolute neutrophil count (ANC) <300/mm3. Doxorubicin, mercaptopurine and methotrexate will be reduced for WBC < 1500/mm3, or if WBC and ANC not increase by at least 2 folds a week after the start date of dexamethasone pulse.

    Reinduction Treatment - This phase of treatment is part of continuation and will be started at weeks 7 and 17 after bone marrow examination confirms complete remission. Doxorubicin and HD-cytarabine will be held if ANC < or equal to 300/mm3 or WBC < 1000/mm3.It is preferable to start HD-cytarabine when WBC > or equal to 1800/mm3 and ANC > 300/mm3 Reinduction treatment will be given twice: weeks 7 to 9 and weeks 17 to 19 for all patients. Intrathecal treatment will be followed by leucovorin rescue (5 mg/m2/dose PO, max 5 mg) at 24 and 30 hours only in patients with prior CNS toxicities or in patients with WBC < 1500/mm3, or ANC < 500/mm3.

    - Reinduction I for Standard/High Risk ALL excluding MLL infants: Dexamethasone 8 mg/m2/day PO (divided t.i.d.) Days 1-8, 15-21. Vincristine 1.5 mg/m2/week IV Days 1, 8, 15 Doxorubicin 30 mg/m2 IV Days 1, 8. PEG-asparaginase 2,500 or 3,500 units/m2 IV Days 1, 15.

    Intrathecal chemotherapy, Methotrexate + hydrocortisone + Ara-C dose age dependent, Day 1.

    - Reinduction II for Standard/High Risk ALL including MLL infants: Dexamethasone 8 mg/m2/day PO (t.i.d.) Days 1-8, 15-21. Vincristine 1.5 mg/m2/week IV Days 1, 8, 15. PEG-asparaginase 2,500 or 3,500 units/m2 IV Days 1, 15. High-dose cytarabine 2 gm/m2 IV q 12 hr Days 15, 16. Intrathecal chemotherapy, dose age dependent, Day 1.

    - Reinduction I for Low-Risk ALL: Dexamethasone 8 mg/m2/day PO (divided t.i.d.) Days 1-8, 15-21. Vincristine 1.5 mg/m2/week IV Days 1, 8, 15. PEG-asparaginase 2,500 or 3,500 units/m2 IV Days 1, 15. Doxorubicin 30 mg/m2/IV Day 1. Intrathecal chemotherapy, dose age dependent, Day 1.

    - Reinduction II for Low-Risk ALL: Dexamethasone 8 mg/m2/day PO (divided t.i.d.) Days 1-8, 15-21. Vincristine 1.5 mg/m2/week IV Days 1, 8, 15. PEG-asparaginase 2,500 or 3,500 units/m2 IV Days 1, 15. Intrathecal chemotherapy, dose age dependent, Day 1.

    - Reinduction I for MLL Infants: Dexamethasone 8 mg/m2/day PO (divided t.i.d.) Days 1-8 and 15-21. Clofarabine 40 mg/m2/day, -hour IV Days 1-5. Etoposide 100 mg/m2/day, 2-hour IV Days 1-5. cyclophosphamide 300 mg/m2/day, 1-hour IV Days 1-5. PEG-asparaginase 2,500 or 3,500 units/m2 IV Days 1, 15. Intrathecal chemotherapy, dose age dependent, on Day 1.

    - Intrathecal Chemotherapy:
    * Triple intrathecal treatment will be given to low-risk cases with CNS-1 status (no identifiable blasts in CSF) on weeks 7, 12, 17, 25, 33, 41, and 49.
    * Triple intrathecal treatment will be given to low-risk cases with CNS-2, traumatic CSF with blasts status, or WBC > 100 x 109/L on weeks 3, 7, 12, 17, 25, 29, 33, 37, 41, 45 and 49.
    * Triple intrathecal treatment will be given to standard/high-risk cases on weeks 7, 12, 17, 25, 29, 33, 37, 41, 45 and 49.
    * Triple intrathecal treatment will be given to other standard/high-risk cases with WBC > or equal to 100 x 109/L, T-cell ALL, t (1;19)/E2A-PBX1, presence of Philadelphia chromosome, MLL rearrangement, hypodiploidy <44, CNS-2 or CNS-3 status, or traumatic lumbar puncture with blasts on weeks 3, 7, 12, 17, 25, 29, 33, 37, 41, 45, 49, 57, 65, 73, 81, 89 and 97

    Treatment (weeks 21 to 29)

    Week Standard/High Risk Low Risk
21. MP + PEG-ASP+Dasatinib MP + MTX
22. MP +Dasatinib MP + MTX
23. MP + PEG-ASP + Dasatinib MP + MTX
24. Cyclo + Ara-C + Dasatinib MP + MTX
25. DEX + VCR + PEG-ASP + Dasatinib MP + DEX + VCR
26. MP + Dasatinib MP + MTX
27. MP + PEG-ASP+Dasatinib MP + MTX
28. Cyclo + Ara-C + Dasatinib MP + MTX
29. DEX + VCR +PEG-ASP + Dasatinib MP + DEX + VCR Dasatinib in Ph+ only

    Treatment (weeks 30 to end of therapy)

    Week Standard/High Risk Low Risk
30. MP + MTX + Dasatinib MP + MTX
31. MP + MTX + Dasatinib MP + MTX
32. Cyclo + Ara-C+Dasatinib MP + MTX
33. DEX + VCR + Dasatinib MP + DEX + VCR
34. MP + MTX + Dasatinib MP + MTX
35. MP + MTX + Dasatinib MP + MTX
36. Cyclo + Ara-C + Dasatinib/MP + MTX
37. DEX + VCR + Dasatinib /MP + DEX + VCR Dasatinib in Ph positive patients only

Drug Dosages, Schedules and Routes for Continuation Therapy from Week 21 to End of Therapy:

Mercaptopurine 75 mg/m2 PO daily for 7 days, Days 1-7. Methotrexate 40 mg/m2 IV or intramuscularly (IM) Day 1. Cyclophosphamide 300 mg/m2 IV, Day 1. Cytarabine 300 mg/m2 IV, Day 1. Dexamethasone 12 mg/m2 (std/high risk) or 8 mg/m2 (low risk) PO daily (divided t.i.d.) for 5 days, Day 1-5 (between week 21 and week 68).Decrease dexamethasone to 6 mg/m2 PO daily (divided t.i.d.) x 5 days,Day 1-5 between week 69 and week 101 for all risk groups.

Vincristine2 mg/m2 IV push (max 2 mg), Day 1 (0.05mg/kg for patients < 1 year or < 10 kg).

PEG-ASP 2,500 vs 3,500 units/m2 IV randomization (until week 30)

Dexamethasone, vincristine, and asparaginase will be given regardless of blood counts, provided that the patient is clinically well. Cyclophosphamide, cytarabine, mercaptopurine and methotrexate will be held if WBC <1000/mm3 or ANC <300/mm3. Mercaptopurine and methotrexate will be reduced for WBC < 1500/mm3, or if WBC and ANC do not increase by at least 2 folds a week after the start date of dexamethasone pulse. Doses of cyclophosphamide and cytarabine may need to be reduced if patient misses 25% of chemotherapy and if the low counts deem to be related to this combination.

The same treatment (weeks 30-37) will be repeated for a total of 5 times, until week 69 (see Section 5.5.3 for intrathecal therapy). After week 69, all patients will receive daily mercaptopurine and weekly methotrexate interrupted with pulses of dexamethasone, vincristine, and mercaptopurine every 4 weeks. The dose of dexamethasone will be decreased to 6 mg/m2 between week 69 and week 101, after which only mercaptopurine and methotrexate will be given. Intrathecal treatment will be given every 8 weeks only to patients at risk of CNS relapse after week 49 and will be discontinued after week 97. Continuation therapy will be discontinued after 120 weeks.

Hematopoietic Stem Cell Transplantation (for patients who meet the criteria of high-risk ALL are candidates for allogeneic hematopoietic stem cell transplantation). However, if the option is declined by the patients or guardians, or the procedure is deemed unsuitable by the attending physician and the principal investigator, the patient will remain on study and continue to receive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a confirmed diagnosis of precursor B-cell or precursor T-cell acute lymphocytic leukemia (ALL) by immunophenotyping
* Participant is less than or equal to 18 years of age
* Limited prior therapy, including systemic glucocorticoids for one week or less, one dose of vincristine, emergency radiation therapy to the mediastinum and one dose of intrathecal chemotherapy. Other circumstances must be cleared by principal investigator (PI) or co-PI.
* Written, informed consent and assent following Institutional Review Board, NCI, FDA, and Office for Human Research Protections (OHRP) Guidelines.

Exclusion Criteria:

* Participants with prior therapy, other than that listed above
* Pregnant or lactating
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Actual)
Dates: Start 2007-10-29 (Actual); Primary Completion 2020-09-26 (Actual); Study Completion 2022-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sima Jeha, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Purvis K, Zhou Y, Karol SE, Rubnitz JE, Ribeiro RC, Lee S, Yang JJ, Bowman WP, Wang L, Dixon SB, Roberts KG, Gao Q, Cheng C, Mullighan CG, Jeha S, Pui CH, Inaba H. Outcomes in patients with ETV6::RUNX1 or high-hyperdiploid B-ALL treated in the St. Jude Total Therapy XV/XVI studies. Blood. 2025 Jan 9;145(2):190-201. doi: 10.1182/blood.2024024936. PMID 39316653
- [Derived] Chang TC, Chen W, Qu C, Cheng Z, Hedges D, Elsayed A, Pounds SB, Shago M, Rabin KR, Raetz EA, Devidas M, Cheng C, Angiolillo A, Baviskar P, Borowitz M, Burke MJ, Carroll A, Carroll WL, Chen IM, Harvey R, Heerema N, Iacobucci I, Wang JR, Jeha S, Larsen E, Mattano L, Maloney K, Pui CH, Ramirez NC, Salzer W, Willman C, Winick N, Wood B, Hunger SP, Wu G, Mullighan CG, Loh ML. Genomic Determinants of Outcome in Acute Lymphoblastic Leukemia. J Clin Oncol. 2024 Oct 10;42(29):3491-3503. doi: 10.1200/JCO.23.02238. Epub 2024 Aug 9. PMID 39121442
- [Derived] Panetta JC, Liu Y, Bottiglieri T, Arning E, Cheng C, Karol SE, Yang JJ, Zhou Y, Inaba H, Pui CH, Jeha S, Relling MV. Pharmacodynamics of cerebrospinal fluid asparagine after asparaginase. Cancer Chemother Pharmacol. 2021 Oct;88(4):655-664. doi: 10.1007/s00280-021-04315-0. Epub 2021 Jun 25. PMID 34170389
- [Derived] Finch ER, Smith CA, Yang W, Liu Y, Kornegay NM, Panetta JC, Crews KR, Molinelli AR, Cheng C, Pei D, Ramsey LB, Karol SE, Inaba H, Sandlund JT, Metzger M, Evans WE, Jeha S, Pui CH, Relling MV. Asparaginase formulation impacts hypertriglyceridemia during therapy for acute lymphoblastic leukemia. Pediatr Blood Cancer. 2020 Jan;67(1):e28040. doi: 10.1002/pbc.28040. Epub 2019 Oct 14. PMID 31612640
- [Derived] Liu Y, Smith CA, Panetta JC, Yang W, Thompson LE, Counts JP, Molinelli AR, Pei D, Kornegay NM, Crews KR, Swanson H, Cheng C, Karol SE, Evans WE, Inaba H, Pui CH, Jeha S, Relling MV. Antibodies Predict Pegaspargase Allergic Reactions and Failure of Rechallenge. J Clin Oncol. 2019 Aug 10;37(23):2051-2061. doi: 10.1200/JCO.18.02439. Epub 2019 Jun 12. PMID 31188727
- [Derived] Hakim H, Dallas R, Wolf J, Tang L, Schultz-Cherry S, Darling V, Johnson C, Karlsson EA, Chang TC, Jeha S, Pui CH, Sun Y, Pounds S, Hayden RT, Tuomanen E, Rosch JW. Gut Microbiome Composition Predicts Infection Risk During Chemotherapy in Children With Acute Lymphoblastic Leukemia. Clin Infect Dis. 2018 Aug 1;67(4):541-548. doi: 10.1093/cid/ciy153. PMID 29518185
- [Derived] Wolf J, Tang L, Flynn PM, Pui CH, Gaur AH, Sun Y, Inaba H, Stewart T, Hayden RT, Hakim H, Jeha S. Levofloxacin Prophylaxis During Induction Therapy for Pediatric Acute Lymphoblastic Leukemia. Clin Infect Dis. 2017 Nov 13;65(11):1790-1798. doi: 10.1093/cid/cix644. PMID 29020310
- [Derived] Bhojwani D, Darbandi R, Pei D, Ramsey LB, Chemaitilly W, Sandlund JT, Cheng C, Pui CH, Relling MV, Jeha S, Metzger ML. Severe hypertriglyceridaemia during therapy for childhood acute lymphoblastic leukaemia. Eur J Cancer. 2014 Oct;50(15):2685-94. doi: 10.1016/j.ejca.2014.06.023. Epub 2014 Jul 30. PMID 25087182
- [Derived] Fernandez CA, Smith C, Yang W, Date M, Bashford D, Larsen E, Bowman WP, Liu C, Ramsey LB, Chang T, Turner V, Loh ML, Raetz EA, Winick NJ, Hunger SP, Carroll WL, Onengut-Gumuscu S, Chen WM, Concannon P, Rich SS, Scheet P, Jeha S, Pui CH, Evans WE, Devidas M, Relling MV. HLA-DRB1*07:01 is associated with a higher risk of asparaginase allergies. Blood. 2014 Aug 21;124(8):1266-76. doi: 10.1182/blood-2014-03-563742. Epub 2014 Jun 26. PMID 24970932
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 29, 2007 and March 26, 2017, 600 patients younger than 19 years of age with newly diagnosed Acute Lymphoblastic Leukemia (ALL) were enrolled.
Pre-assignment Details: Two (2) were later found ineligible and excluded. Of the 598 eligible patients, 414 patients were randomized to the two treatment arms, 184 were not randomized for various reasons:
  * Not Eligible for Randomization (n=41)
    * Death (n=5)
    * Transplant (n=13)
    * Withdrawal of Consent (n=3)
    * Down's Syndrome (n=12)
    * Poor Organ Function (n=8)
  * Parent/Patient Decision (n=70)
  * Attending Physician Decision (n=4)
  * Enrollment after Completion of Randomization (n=69)
Groups:
- PEG 3500 Units/m^2: Patients randomized on the first day of continuation phase to receive 3500 units/m^2 dose of PEG-asparaginase
- PEG 2500 Units/m^2: Patients randomized on the first day of continuation phase to receive 2,500 units/m^2 dose of PEG-asparaginase
- Not Randomized: Patients who came off study prior to randomization
Period: Overall Study
Arm/Group | PEG 3500 Units/m^2 | PEG 2500 Units/m^2 | Not Randomized
Started | 206 | 208 | 184
Completed | 194 | 188 | 133
Not Completed | 12 | 20 | 51
Not completed — Death | 1 | 4 | 13
Not completed — Physician Decision | 0 | 0 | 4
Not completed — Bone Marrow (BM) or Extramedullary Relapse | 3 | 4 | 4
Not completed — Failure to achieve Complete Remission (CR) | 1 | 0 | 1
Not completed — Participant/Family Withdraw | 2 | 3 | 5
Not completed — Second Malignancy | 1 | 0 | 0
Not completed — Transplant | 3 | 3 | 18
Not completed — Unacceptable Toxicity | 1 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEG 3500 Units/m^2 | PEG 2500 Units/m^2 | Not Randomized | Total
Number analyzed (Participants) | 206 | 208 | 184 | 598
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.13 (4.78) | 7.04 (4.73) | 7.75 (5.04) | 7.29 (4.85)
Age, Customized [Count of Participants; unit: Participants]
  <1 year | 5 | 3 | 4 | 12
  1-10 years | 152 | 160 | 131 | 443
  >10 years | 49 | 45 | 49 | 143
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 85 | 72 | 248
  Male | 115 | 123 | 112 | 350
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Cuban | 1 | 0 | 0 | 1
  Mexican/Chicano | 7 | 5 | 7 | 19
  NOS Spanish,Hispanic,Latino | 13 | 14 | 13 | 40
  Non Spanish speaking, Non Hispanic | 182 | 187 | 161 | 530
  Puerto Rican | 0 | 0 | 1 | 1
  South or Central Amercian | 2 | 0 | 2 | 4
  Unknown | 1 | 2 | 0 | 3
  White | 154 | 167 | 143 | 464
  Black | 34 | 29 | 25 | 88
  Other | 18 | 12 | 16 | 46
Region of Enrollment [Number; unit: participants]
  United States | 206 | 208 | 184 | 598

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Continuous Complete Remission of Patients Receiving High-dose and Conventional Dose PEG-asparaginase.
Description: The primary objective of this study is to compare the distributions of continuous complete remission of patients randomized on the first day of the continuation phase to receive a higher dose of PEG-asparaginase or to receive the conventional dose (2,500 units/m2).
  The randomization will occur on the starting day of the continuation phase, at which time all information necessary for performing the randomization should be available. In the rare case that immunophenotype and/or Day-15 MRD is not available, we will make the following assumptions: If immunophenotype is unknown at the time the randomization is to be executed, then it will be assumed B-lineage. If Day-15 MRD is unknown at the time of randomization, then it will be assumed negative (<0.01%). Past experience indicate that few patients will fall into these unknown categories.
Time Frame: 3.5 years after the last enrollment up to 12.5 years
Population: Per protocol, the comparison was between the two randomization arms.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG 3500 Units/m^2 | PEG 2500 Units/m^2
Number analyzed (Participants) | 206 | 208
Percentage of participants | 91.6 [87.7 to 95.5] | 90.7 [86.6 to 94.8]
Statistical Analysis 1: Comparison: PEG 3500 Units/m^2 vs PEG 2500 Units/m^2; Test type: Superiority; p = 0.778, Cochran-Mantel-Haenszel

2. Secondary Outcome: Probability of Event-free Survival
Description: To estimate the event-free survival of children with ALL who are treated with risk-directed therapy and to compare the EFS results of TOTXVI with that of TOTXV (NCT00137111).
  EFS will be measured from the date of complete response to the date of initial failure for patients who fail. Failure includes the traditional endpoints of failure to achieve a complete remission, relapse in any site, secondary malignancy, and death during induction or remission. EFS time will be measured to the date of last contact for patients who are failure free at the time of analysis. The EFS time is defined to be zero (0) for patients who die during induction therapy or fail to achieve a complete remission.
Time Frame: For Total XVI: 3.5 years after the last enrollment, up to approximately 13.5 years For Total XV: patients are followed continuously, up to 20.5 years
Population: Per protocol this objective is to study whether intensifying induction will result in improved outcome compared to TOTXV. All eligible patients entered on TOTXVI will be included in these analyses, as appropriate. Infants will be excluded from the Total XVI for comparisons with TOTXV as only children at least one year of age at diagnosis were treated on Total XV.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- TOTXVI PEG 3500: Patients randomized on the first day of continuation phase to receive 3500 units/m^2 dose of PEG-asparaginase
- TOTXVI PEG 2500: Patients randomized on the first day of continuation phase to receive 2,500 units/m^2 dose of PEG-asparaginase
- TOTXVI Not Randomized: Patients who came off study prior to randomization
- All Eligible Patients in TOTXV: All 498 eligible children with ALL who are treated with risk-directed therapy.
Arm/Group | TOTXVI PEG 3500 | TOTXVI PEG 2500 | TOTXVI Not Randomized | All Eligible Patients in TOTXV
Number analyzed (Participants) | 201 | 205 | 180 | 498
Percentage of participants | 92.4 [88.7 to 96.1] | 91.1 [87.0 to 95.2] | 86.3 [78.9 to 93.7] | 87.1 [84.2 to 90.0]

3. Secondary Outcome: Probability of Overall Survival
Description: To estimate the overall survival of children with ALL who are treated with risk-directed therapy and to compare the EFS results of TOTXVI with that of TOTXV.
Time Frame: as for outcome 2
Population: All eligible patients entered on TOTXVI will be included in these analyses, as appropriate. Infants will be excluded from the Total XVI for comparisons with TOTXV as only children at least one year of age at diagnosis were treated on Total XV.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- TOTVI Not Randomized: Patients who came off study prior to randomization
- All Eligible Patients in TOTXV: All eligible children with ALL who are treated with risk-directed therapy.
Arm/Group | TOTXVI PEG 3500 | TOTXVI PEG 2500 | TOTVI Not Randomized | All Eligible Patients in TOTXV
Number analyzed (Participants) | 201 | 205 | 180 | 498
Percentage of participants | 97.5 [95.3 to 99.7] | 95.6 [92.7 to 98.5] | 90.8 [84.7 to 96.9] | 93.5 [91.3 to 95.7]

4. Secondary Outcome: Proportion of Participants With Minimal Residual Disease (MRD) on the 15th Day of Remission Induction ≥ 5%
Description: To study whether intensifying induction, including fractionated cyclophosphamide and thioguanine, in patients with day 15 MRD ≥ 5% will result in improved leukemia cytoreduction in this subgroup compared to therapy followed in the TOTXV protocol.
Time Frame: Middle of remission induction, Day 15 in Total XVI and Day 19 in Total XV
Population: The analysis will compare the proportion of TOTXV patients who had Day-19 MRD≥5% with the proportion of patients on TOTXVI with Day-15 MRD≥5%.
Measure: Count of Participants; unit: Participants
Groups:
- All Eligible Patients in TOTXV: Eligible Patients in TOTXV
Arm/Group | TOTXVI PEG 3500 | TOTXVI PEG 2500 | TOTXVI Not Randomized | All Eligible Patients in TOTXV
Number analyzed (Participants) | 203 | 206 | 183 | 488
Participants | 22 | 26 | 31 | 55

5. Secondary Outcome: Proportion of Participants With Minimal Residual Disease (MRD) at End of Remission Induction ≥ 0.01%
Description: as for outcome 4
Time Frame: End of remission induction; day 42 in Total XVI and day 46 in Total XV
Population: We will compare the proportion of patients with Day-15 MRD≥5% on TOTXVI who are Day-42 MRD positive with the proportion of Day-46 MRD positives in the corresponding subgroup in TOTXV by Fisher's exact test.
Measure: Count of Participants; unit: Participants
Groups:
- All Eligible Patients in TOTXV: Day 15 MRD > or equal to 5% in Total XV
Arm/Group | TOTXVI PEG 3500 | TOTXVI PEG 2500 | TOTXVI Not Randomized | All Eligible Patients in TOTXV
Number analyzed (Participants) | 22 | 26 | 30 | 54
Participants | 7 | 12 | 20 | 44

6. Secondary Outcome: Probability of CNS Relapse
Description: To assess whether intensification of CNS-directed intrathecal and systemic chemotherapy will improve outcome in patients at high-risk of CNS relapse.
Time Frame: as for outcome 2
Population: Patients with features associated with increased risk for CNS relapse in Total XVI and Total XV.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All Eligible Patients in TOTXV: Patients with features associated with increased risk for CNS relapse in Total XV
Arm/Group | TOTXVI PEG 3500 | TOTXVI PEG 2500 | TOTXVI Not Randomized | All Eligible Patients in TOTXV
Number analyzed (Participants) | 121 | 125 | 113 | 248
Percentage of participants | 0.8 [0.0 to 2.5] | 1.8 [0.0 to 4.3] | 2.7 [0.0 to 5.7] | 5.7 [2.8 to 8.6]

ADVERSE EVENTS:
Time Frame: Through 1 month after therapy completion, approximately 25 months
Description: Systemic assessment was used for collection of adverse events including:
  * Real time reporting of significant events by treating team
  * Regular communication with families and close monitoring of medical records, laboratory results, and imaging by dedicated research nurse (daily for inpatient setting and weekly for outpatient setting)
  * Biweekly review of AEs by PI and treating team for accuracy and completion
Arm/Group | PEG 3500 Units/m^2 | PEG 2500 Units/m^2 | Not Randomized
All-Cause Mortality (participants affected / at risk) | 9/206 | 15/208 | 22/184
Serious Adverse Events (participants affected / at risk) | 0/206 | 0/208 | 2/184
Other Adverse Events (participants affected / at risk) | 206/206 | 208/208 | 184/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG 3500 Units/m^2 (N=206) | PEG 2500 Units/m^2 (N=208) | Not Randomized (N=184)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Infection, Blood (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG 3500 Units/m^2 (N=206) | PEG 2500 Units/m^2 (N=208) | Not Randomized (N=184)
Allergic reaction to Asparaginase (Injury, poisoning and procedural complications) | 28 (36) | 30 (35) | 18 (20)
Hypertension (Vascular disorders) | 50 (58) | 47 (56) | 58 (66)
Hypotension (Vascular disorders) | 16 (17) | 19 (23) | 10 (13)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 156 (395) | 147 (381) | 116 (283)
Dehydration (Metabolism and nutrition disorders) | 19 (22) | 10 (11) | 13 (14)
Diarrhea (Gastrointestinal disorders) | 17 (19) | 12 (13) | 11 (12)
Mucositis/stomatitis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 47 (64) | 63 (78) | 36 (46)
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 19 (25) | 25 (37) | 19 (21)
Vomiting (Gastrointestinal disorders) | 16 (17) | 16 (18) | 17 (18)
Pancreatitis (Gastrointestinal disorders) | 13 (17) | 19 (24) | 28 (44)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 83 (168) | 61 (103) | 55 (113)
Febrile neutropenia (Blood and lymphatic system disorders) | 163 (392) | 160 (404) | 124 (239) — Fever of unknown origin without clinically or microbiologically documented infection (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Infection, Blood (Infections and infestations) | 38 (49) | 48 (66) | 45 (51) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection, Catheter-related (Infections and infestations) | 14 (16) | 17 (22) | 8 (8) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection, Lip/perioral (Infections and infestations) | 9 (13) | 17 (23) | 8 (10) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection, Lung (pneumonia) (Infections and infestations) | 37 (42) | 47 (63) | 22 (28) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection, Middle ear (otitis media) (Infections and infestations) | 30 (36) | 38 (48) | 22 (28) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection, Oral cavity-gums (gingivitis) (Infections and infestations) | 32 (41) | 35 (55) | 27 (36) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection, Rectum (Infections and infestations) | 7 (7) | 15 (15) | 11 (11) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection, Sinus (Infections and infestations) | 21 (25) | 23 (25) | 6 (8) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection, Skin (cellulitis) (Infections and infestations) | 42 (52) | 41 (47) | 39 (49) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection, Upper airway NOS (Infections and infestations) | 92 (129) | 110 (186) | 85 (143) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection, Urinary tract NOS (Infections and infestations) | 11 (15) | 14 (22) | 7 (8) — Documented clinically or microbiologically with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection with normal ANC or Grade 1 or 2 neutrophils, Blood (Infections and infestations) | 23 (33) | 26 (27) | 20 (25)
Infection with normal ANC or Grade 1 or 2 neutrophils, Catheter-related (Infections and infestations) | 16 (18) | 8 (8) | 8 (8)
Infection with normal ANC or Grade 1 or 2 neutrophils, Conjunctiva (Infections and infestations) | 20 (22) | 18 (23) | 15 (16)
Infection with normal ANC or Grade 1 or 2 neutrophils, External ear (otitis externa) (Infections and infestations) | 11 (13) | 13 (15) | 7 (8)
Infection with normal ANC or Grade 1 or 2 neutrophils, Lip/perioral (Infections and infestations) | 35 (74) | 28 (56) | 14 (32)
Infection with normal ANC or Grade 1 or 2 neutrophils, Lung (pneumonia) (Infections and infestations) | 49 (57) | 46 (50) | 30 (38)
Infection with normal ANC or Grade 1 or 2 neutrophils, Middle ear (otitis media) (Infections and infestations) | 84 (197) | 80 (146) | 56 (117)
Infection with normal ANC or Grade 1 or 2 neutrophils, Oral cavity-gums (gingivitis) (Infections and infestations) | 50 (82) | 48 (92) | 47 (96)
Infection with normal ANC or Grade 1 or 2 neutrophils, Sinus (Infections and infestations) | 66 (136) | 51 (78) | 29 (46)
Infection with normal ANC or Grade 1 or 2 neutrophils, Skin (cellulitis) (Infections and infestations) | 91 (167) | 80 (127) | 70 (116)
Infection with normal ANC or Grade 1 or 2 neutrophils, Ungual (nails) (Infections and infestations) | 19 (28) | 6 (6) | 9 (12)
Infection with normal ANC or Grade 1 or 2 neutrophils, Upper airway NOS (Infections and infestations) | 133 (306) | 136 (301) | 105 (262)
Infection with normal ANC or Grade 1 or 2 neutrophils, Urinary tract NOS (Infections and infestations) | 25 (34) | 23 (33) | 16 (32)
Infection with normal ANC or Grade 1 or 2 neutrophils, Vagina (Infections and infestations) | 11 (21) | 13 (15) | 8 (15)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 32 (39) | 30 (47) | 29 (41)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 22 (25) | 25 (34) | 21 (23)
Bilirubin (hyperbilirubinemia) (Investigations) | 11 (12) | 14 (17) | 19 (24)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 22 (35) | 23 (30) | 25 (38)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 19 (22) | 22 (30) | 13 (13)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 19 (23) | 18 (19) | 17 (18)
Fracture (Injury, poisoning and procedural complications) | 19 (24) | 25 (29) | 21 (23)
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 85 (188) | 79 (189) | 57 (152)
Neuropathy: motor (Nervous system disorders) | 53 (53) | 54 (57) | 56 (58)
Seizure (Nervous system disorders) | 14 (14) | 9 (10) | 12 (13)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 36 (45) | 38 (53) | 36 (42)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 10 (10) | 9 (9)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 25 (25) | 36 (36) | 24 (24)
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 8 (9) | 12 (12) | 12 (12)
Pain, Abdomen NOS (Gastrointestinal disorders) | 43 (53) | 32 (40) | 22 (28)
Pain, Back (Musculoskeletal and connective tissue disorders) | 22 (26) | 14 (19) | 12 (12)
Pain, Extremity-limb (Musculoskeletal and connective tissue disorders) | 11 (11) | 17 (18) | 4 (4)
Pain, Head/headache (Nervous system disorders) | 22 (27) | 20 (24) | 18 (19)
Pain, Neuralgia/peripheral nerve (Nervous system disorders) | 155 (221) | 160 (218) | 128 (157)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT00549848/Prot_SAP_000.pdf